CLINICAL TRIAL: NCT05661240
Title: Phase Ⅱ/Ⅲ Clinical Study of Tumor Treating Fields（EFE-P100） Combined With Docetaxel in the Treatment of Stage IV Non-small Cell Lung Cancer Patients With Disease Progression After Platinum-based Chemotherapy and Anti-programmed Death 1(PD-1)/Programmed Cell Death-Ligand 1(PD-L1) Antibody Treatment
Brief Title: Phase Ⅱ/Ⅲ Clinical Study of Tumor Treating Fields （EFE-P100）Combined With Docetaxel in the Treatment of Stage IV Non-small Cell Lung Cancer Patients With Disease Progression After Platinum-based Chemotherapy and Anti-programmed Death 1（PD-1)/Programmed Cell Death-Ligand 1(PD-L1) Antibody Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Healthy Life Innovation Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100-NSCLC2
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumor treating fields combined with docetaxel injection (Experimental): Medical device：Tumor treating fields（EFE-P100） Tumor treating fields（EFE-P100）will be used each day. Drug: docetaxel each cycle is 21 days，docetaxel will be administered intravenously，75 mg/m2 on the first day of each cycle.
  Interventions: Device: Tumor treating fields（EFE-P100）; Drug: Docetaxel injection
- docetaxel injection (Active Comparator): Drug: docetaxel each cycle is 21 days，docetaxel will be administered intravenously，75 mg/m2 on the first day of each cycle.
  Interventions: Drug: Docetaxel injection

INTERVENTIONS:
Device: Tumor treating fields（EFE-P100） — Device: Tumor treating fields（EFE-P100） Subjects will use EFE-P100 until disease progression or for a maximum of 24 months.
  Arms: Tumor treating fields combined with docetaxel injection
Drug: Docetaxel injection — Drug: Docetaxel injection Subjects will receive Docetaxel injection until disease progression or for a maximum of 24 months.

SUMMARY:
The tumor treating fields（EFE-P100）generates alternating electric field during operation, and the tumor treating fields（EFE-P100）has a specific frequency and a specific field intensity. The tumor treating fields（EFE-P100）patch acts on the corresponding part of the patient and prevents the mitosis of tumor cells. This study was divided into two phases including phase II and phase III clinical trials. The main purpose of phase II clinical trial is to evaluate the safety of tumor treating fields（EFE-P100） combined with docetaxel injection in the second-line treatment of stage IV non-small Cell Lung Cancer (NSCLC) patients who failed after platinum-containing chemotherapy and anti-programmed Death 1（PD-1)/Programmed Cell Death-Ligand 1(PD-L1) antibody treatment. The main purpose of phase III clinical trial is to compare the efficacy of tumor treating fields（EFE-P100） combined with docetaxel injection and docetaxel injection alone in the second-line treatment of stage IV non-small cell lung cancer (NSCLC) patients who failed after platinum-containing chemotherapy and anti-programmed Death 1（PD-1)/Programmed Cell Death-Ligand 1(PD-L1) antibody treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80, both sexes;
2. Expected survival time ≥3 months;
3. Non-small cell lung cancer was confirmed histologically or cytologically and classified as stage IV NSCLC according to the American Joint Committee on Cancer（AJCC）of eighth edition.
4. Imaging progression (according to RECIST V1.1 criteria) or clinical progression during previous anti-PD - (L) 1 antibody and platinum-containing therapy or after treatment; - Neoadjuvant or adjuvant therapy, such as disease recurrence or progression ≤6 months after the end of treatment, counted as first-line treatment; - Prior treatment with at least 2 cycles of anti-PD - (L) 1 antibody, allowed as a single agent or in combination with platinum-based chemotherapy.
5. At least one measurable or evaluable lesion according to RECIST version 1.1;
6. ECOG 0-1;
7. Concomitant Adverse Event（AE） after previous treatment should return to normal level or Common Terminology Criteria for Adverse Events（CTCAE） grade 1;
8. Voluntarily sign informed consent.

Exclusion Criteria:

1. Epidermal growth factor receptor（EGFR）-activating mutations or Anaplastic Lymphoma Kinase（ALK） fusion gene was positive; However, if squamous non-small cell lung cancer has not been tested before, it can no longer be tested and allowed to be enrolled.
2. Untreated brain metastases, or with meningeal metastases, spinal cord compression, etc. Patients who had received previous treatment for brain metastases and were asymptomatic if they had been stable for at least 4 weeks on imaging before randomization and had stopped systemic hormone therapy (dose >10mg/ day prednisone or other equivalent hormone) for more than 2 weeks were eligible.
3. Severe bone injury due to bone metastases, including severe bone pain that is poorly controlled, pathologic fractures of major sites that have occurred within the last 6 months or are expected to occur in the near future.
4. Previous docetaxel therapy or docetaxel-containing combination therapy;
5. There are contraindications to docetaxel treatment or a known severe allergy to docetaxel;
6. A history of diagnosis of a tumor other than small-cell lung cancer and antitumor therapy within 5 years prior to enrollment, excluding treated stage I prostate cancer, cervical or uterine cancer in situ, breast cancer in situ, and non-melanoma skin cancer;
7. Abnormal bone marrow, heart, liver and kidney function: A. Neutrophil count <1.5×109/L, platelet count <100×109/L, hemoglobin <90 g/L; TBiL> upper normal value (ULN); AST and/or ALT>2.5×ULN; ALP>2.5×ULN (>5×ULN if bone metastases are present); C. Serum creatinine >1.5×ULN; Creatinine clearance rate <50 mL/min;
8. A history of severe cardiovascular disease, including second/third degree heart block; Severe ischemic heart disease; Poor control of hypertension; New York Heart Association (NYHA) class II or worse congestive heart failure (mild physical activity limitation; Comfortable at rest, but normal activities can cause fatigue, palpitations, or difficulty breathing);
9. Patients who required systemic corticosteroid (other corticosteroid at a dose of more than 10mg prednisone per day or an equivalent physiologic dose) or other immunosuppressive agents within 14 days prior to enrollment or during the study period were eligible for enrollment if: A. The use of topical or inhaled glucocorticoids is permitted; B. Allow short-term (≤7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases;
10. If she had severe infection before the first treatment, the investigator judged that she was not suitable to participate in this study.
11. A history of human immunodeficiency virus (HIV) infection (known HIV1/2 antibody positive);
12. The presence of active hepatitis B, active hepatitis C, or other active infections that the investigator determines may affect the patient's treatment;
13. There is a definite history of neurological or psychiatric disorders (e.g., epilepsy, dementia) or drug use or alcohol abuse within the last year that may affect trial compliance;
14. Symptomatic ascites, pleural effusion, pericardial effusion, etc., except those who are stable after clinical treatment (including therapeutic puncture);
15. Infection, ulceration and unhealed wound on the skin where the electrode is applied;
16. Currently participating in other antitumor therapy clinical trials;
17. Implantable electronic medical devices, such as pacemakers;
18. Chest and abdomen have implanted metal materials of medical instruments, such as bone nails;
19. Allergic to conductive hydrogels or medical adhesives;
20. Pregnant or trying to become pregnant or breastfeeding;
21. Poor compliance or other factors as judged by the investigator were not appropriate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2024-05-25 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with Tumor Treating Fields（EFE-P100） and Docetaxel until the first documentation of disease progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | The whole study period，an average of 2 year
  Will be defined as the incidence, frequency and severity of adverse events (AEs) noted in patients treated with study treatments
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1.
Overall survival (OS) | up to 12 months after the last study treatment
  From date of enrollment until the date of death from any cause
12-month OS rate | 12 months
  12-month Overall survival rate
Progression Free Survival rate at 6 months | 6 months
  The analysis will be estimated proportions of patients who are progression-free at 6 months based on the RECIST 1.1 criteria following the time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Zhou, Principal Investigator — MD
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No